CLINICAL TRIAL: NCT00440830
Title: Study to Determine Whether the Use of a Nicotine Patch During the Day of Surgery Improves Postoperative Pain and Reduces Opioid Requirement
Brief Title: Nicotine Patch as an Analgesic Adjuvant After Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AAAB5945
Record Dates: First submitted 2007-02-26; First posted 2007-02-27 (Estimated); Results first posted 2010-10-27 (Estimated); Last update posted 2021-10-21 (Actual); Status verified 2021-09

CONDITIONS: Pain
Keywords: acute pain; nicotine; nausea; sedation
MeSH Terms: conditions — Pain; Acute Pain; Nausea | interventions — Tobacco Use Cessation Devices; Nicotine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Smokers-nicotine (Experimental): Smokers who were treated with nicotine
  Interventions: Drug: nicotine patch
- Nonsmokers-nicotine (Experimental): Nonsmokers who were treated with nicotine
  Interventions: Drug: nicotine patch
- Smokers-placebo (Placebo Comparator): Smokers who were treated with placebo
  Interventions: Drug: placebo
- Nonsmokers-placebo (Placebo Comparator): Nonsmokers who were treated with placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: nicotine patch — nicotine patch (0,5,10 or 15mg/day) applied to smokers
  Other Names: nicotrol
  Arms: Smokers-nicotine
Drug: nicotine patch — nicotine patch (0,5,10,or 15mg/day) applied to nonsmokers
  Other Names: nicotrol
  Arms: Nonsmokers-nicotine
Drug: placebo — placebo patch applied to smokers
  Arms: Smokers-placebo
Drug: placebo — placebo patch applied to nonsmokers
  Arms: Nonsmokers-placebo

SUMMARY:
Effect of nicotine patch as an adjutant for acute pain after surgery.

DETAILED DESCRIPTION:
This is a dose finding trial for nicotine patches as analgesics. Doses used are 5mg/ 10mg/ 15mg or placebo. Primary outcome variable is reported pain score (VAS), secondary is morphine PCA utilization, nausea, sedation, and hemodynamic changes.

ELIGIBILITY:
Inclusion Criteria:

* Adult ASA 1-2

Exclusion Criteria:

* Cardiovascular disease
* Former smoker
* Pregnant
* Nursing
* Asthma

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2005-12; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Flood, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center / New York Presbyterian, New York, New York, United States

REFERENCES:
- [Result] Olson LC, Hong D, Conell-Price JS, Cheng S, Flood P. A transdermal nicotine patch is not effective for postoperative pain management in smokers: a pilot dose-ranging study. Anesth Analg. 2009 Dec;109(6):1987-91. doi: 10.1213/ANE.0b013e3181bd1612. PMID 19923530
- [Result] Hong D, Conell-Price J, Cheng S, Flood P. Transdermal nicotine patch for postoperative pain management: a pilot dose-ranging study. Anesth Analg. 2008 Sep;107(3):1005-10. doi: 10.1213/ane.0b013e318163204f. PMID 18713921

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This prospective, double-blind trial was approved by the IRB at Columbia University Medical Center. All patients signed written informed consent before surgery.
Groups:
- Smokers-nicotine: Nicotine patch (0,5,10 or 15mg/day) was applied to hairless skin away from the surgical site 1 hour before induction of smoking patients.
- Smokers-placebo: Placebo patch was applied to hairless skin away from the surgical site 1 hour before induction of smoking patients.
- Non-smokers-nicotine: Nicotine patch (0,5,10 or 15mg/day) was applied to hairless skin away from the surgical site 1 hour before induction of nonsmoking patients.
- Non-smokers-placebo: Placebo patch was applied to hairless skin away from the surgical site 1 hour before induction of nonsmoking patients.
Period: Overall Study
Arm/Group | Smokers-nicotine | Smokers-placebo | Non-smokers-nicotine | Non-smokers-placebo
Started | 20 | 8 | 30 | 10
Completed | 20 | 8 | 30 | 10
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Smokers-nicotine | Smokers-placebo | Non-smokers-nicotine | Non-smokers-placebo | Total
Number analyzed (Participants) | 20 | 8 | 30 | 10 | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 8 | 30 | 10 | 68
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (2) | 43 (4) | 48 (3) | 52 (4) | 47 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 5 | 15 | 5 | 42
  Male | 3 | 3 | 15 | 5 | 26
Region of Enrollment [Number; unit: participants]
  United States | 20 | 8 | 30 | 10 | 68

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Pain Score One Hour After Surgery
Description: Postoperative pain reported after the first hour using a standard numerical rating scale (NRS) with 0=no pain and 10=worst pain imaginable.
Time Frame: 1 hour after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Smokers-nicotine | Smokers-placebo | Non-smokers-nicotine | Non-smokers-placebo
Number analyzed (Participants) | 20 | 8 | 30 | 10
score on a scale | 5.78 (1.80) | 5.17 (1.94) | 4.32 (1.78) | 5.60 (1.51)

2. Primary Outcome: Postoperative Pain Score Five Days After Surgery
Description: Postoperative pain reported after five days using a standard numerical rating scale (NRS) with 0=no pain and 10=worst pain imaginable.
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Smokers-nicotine | Smokers-placebo | Non-smokers-nicotine | Non-smokers-placebo
Number analyzed (Participants) | 20 | 8 | 30 | 10
score on a scale | 2.24 (2.36) | 3.25 (2.31) | 1.38 (1.08) | 2.70 (1.49)

3. Secondary Outcome: Nausea Assessment by Patient
Description: Nausea scale range: 0=none and 10=the worst, ordinal.
Time Frame: 1 hour after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Smokers-nicotine | Nonsmokers-nicotine | Smokers-placebo | Nonsmokers-placebo
Number analyzed (Participants) | 20 | 30 | 8 | 10
score on a scale | 0 (0) | 2.1 (1.0) | 0 (0) | 2.4 (2.0)

4. Secondary Outcome: Pain Medication Used
Description: Pain medication used after surgery in morphine equivalents
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: Morphine equivalents
Arm/Group | Smokers-nicotine | Smokers-placebo | Non-smokers-nicotine | Non-smokers-placebo
Number analyzed (Participants) | 20 | 8 | 30 | 10
Morphine equivalents | 75.2 (10.7) | 82.0 (22.9) | 41.9 (11.2) | 35.7 (10.5)

5. Secondary Outcome: Systolic Blood Pressure
Description: Systolic blood pressure reported in Millimeters of Mercury (mmHg)
Time Frame: 1 hour after surgery
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury (mmHg)
Arm/Group | Smokers-nicotine | Smokers-placebo | Non-smokers-nicotine | Non-smokers-placebo
Number analyzed (Participants) | 20 | 8 | 30 | 10
Millimeters of Mercury (mmHg) | 131 (21) | 127 (28) | 130 (11) | 136 (21)

6. Secondary Outcome: Diastolic Blood Pressure
Description: Diastolic blood pressure reported in Millimeters of Mercury (mmHg)
Time Frame: 1 hour after surgery
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury (mmHg)
Arm/Group | Smokers-nicotine | Smokers-placebo | Non-smokers-nicotine | Non-smokers-placebo
Number analyzed (Participants) | 20 | 8 | 30 | 10
Millimeters of Mercury (mmHg) | 66 (10.4) | 80 (12) | 72 (23) | 65 (28)

7. Secondary Outcome: Heart Rate
Description: Heart rate reported in Beats per minute (BPM)
Time Frame: 1 hour after surgery
Measure: Mean (Standard Deviation); unit: Beats per minute (BPM)
Arm/Group | Smokers-nicotine | Smokers-placebo | Non-smokers-nicotine | Non-smokers-placebo
Number analyzed (Participants) | 20 | 8 | 30 | 10
Beats per minute (BPM) | 74 (12) | 83 (16) | 72 (11) | 78 (14)

8. Other Pre Specified Outcome: Sedation Level
Description: Sedation may be monitored for the first hour, at the time of other data collection.
Time Frame: 1 hour after surgery
Population: Data was not collected or analyzed for this measure.
Arm/Group | Smokers-nicotine | Nonsmokers-nicotine | Smokers-placebo | Nonsmokers-placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Smokers-nicotine | Smokers-placebo | Non-smokers-nicotine | Non-smokers-placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/8 | 0/30 | 0/10
Other Adverse Events (participants affected / at risk) | 0/20 | 0/8 | 0/30 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes